CLINICAL TRIAL: NCT00057447
Title: Phase I/II Study of the Safety of Subcutaneous Interferon Gamma-1b Combined With Rituximab in Patients With Low Grade/Follicular Non-Hodgkin's Lymphoma
Brief Title: Safety of Interferon Gamma-1b With Rituximab in Non-Hodgkin's Lymphoma Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: administrative reasons
Sponsor: InterMune (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GINHL-001
Record Dates: First submitted 2003-04-01; First posted 2003-04-03 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — interferon gamma-1b; Rituximab

INTERVENTIONS:
Drug: Interferon Gamma-1b — 100 or 200 mcg, SQ, 3x per week
Drug: Rituximab — 375 mg per square meters, IV, 1x per week

SUMMARY:
Evaluate the safety and efficacy of the dosing schedule of subcutaneous interferon gamma-1b (IFN g-1b) administered 3 times per week with Rituximab for 4 weeks, in patients with progressive or relapsed low-grade Non-Hodgkin's Lymphoma (NHL)

International study with sites in the Czech Republic and Poland

ELIGIBILITY:
* Relapsed or progressive low-grade/follicular NHL who are candidates for rituximab therapy
* Patients who were on other therapy including CHOP or radiation
* Previous therapy must have concluded 30 days prior to enrollment
* Demonstrable CD20-positive tumor population in lymph nodes or bone marrow

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-03; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
time to complete response (disappearance of all detectable clinical and radiographic evidenc of disease, and regression of lymph nodes) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Williamson Bradford, MD, Study Director — InterMune
Locations (1):
- Intermune Inc, Brisbane, California, United States